CLINICAL TRIAL: NCT00683280
Title: Contingency Management and Pharmacotherapy for Smoking Cessation
Acronym: Donaghue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-035-3; DF 07-028 (Other Grant/Funding Number: The Ethel Donaghue Center for Translating Research into Practice and Policy)
Record Dates: First submitted 2008-05-14; First posted 2008-05-23 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Cigarette Smoking
Keywords: Contingency Management; Cigarette Smoking Cessation; varenicline
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Medication (varenicline) for 12 weeks (Day 1 through 84) and brief counseling based on public health service guidelines for 5 weeks (Day 1 through 35).
  Interventions: Other: Standard of Care
- Standard of Care plus Contingency Management (Experimental): Medication (varenicline) for 12 weeks (Day 1 through 84), brief counseling based on public health service guidelines for 5 weeks (Day 1 through 35), plus prize-based contingency management for carbon monoxide samples and urinary cotinine samples that meet smoking abstinence criteria.
  Interventions: Behavioral: contingency management; Other: Standard of Care

INTERVENTIONS:
Behavioral: contingency management — Prize-based contingency management, with the opportunity to earn prizes for expired carbon monoxide levels reading 6ppm or less and urinary cotinine levels reading 30ng/ml or less for 4 weeks.
  Arms: Standard of Care plus Contingency Management
Other: Standard of Care — varenicline (smoking cessation medication) 0.5mg po daily Days 1-3, 0.5mg po twice daily Days 4-7, 1.0 mg po twice daily Days 8-84.
Other: Standard of Care — Twice weekly brief counseling based on public health service guidelines for quitting smoking.

SUMMARY:
In total, 70 smokers will be randomized to: standard of care smoking cessation medication varenicline alone (an FDA-approved smoking cessation medication) or varenicline plus contingency management (CM) (a behavioral procedure with rewards for target behaviors, like smoking abstinence). Patients in both conditions will receive varenicline for 12 weeks with standard smoking cessation therapy and regular breath and urine sample monitoring for smoking. Patients assigned to CM will earn chances to win prizes for each breath sample that tests negative for smoking, and urine samples that test negative for smoking will result in even greater chances for prizes. More CM patients are expected to achieve and maintain abstinence than patients receiving varenicline alone.

ELIGIBILITY:
Inclusion Criteria:

* smoke >10 cigarettes/day, with no abstinent period exceeding 3 months in past year
* expired CO of >8 ppm
* self-reported desire to stop smoking
* >18 years of age
* resting systolic BP<160 mmHg and diastolic BP<100 mmHg and otherwise in good health
* if on antihypertensive medication, have not changed medications in the past month and do not intend to change in next 3 months
* English speaking

Exclusion Criteria:

* receipt of smoking cessation treatment (behavioral or pharmacological) in past month
* serious or unstable medical disease in past 6 months, including myocardial infarction, cancer, congestive heart failure, kidney failure, stroke, or seizures
* evidence or history of allergic reactions contraindicating varenicline or clinically significant laboratory or electrocardiographic (ECG) abnormalities
* breastfeeding, pregnant or not using effective contraception if a woman of childbearing potential
* arm circumference of >42 cm
* serious psychiatric illness in past 6 months (e.g., schizophrenia, psychosis, suicide risk, drug or alcohol dependence other than nicotine)
* use of tobacco containing products other than cigarettes in past month and do not agree to abstain from use of these products during study participation
* ongoing use of any of the following medications: nicotine replacement therapies, monoamine oxidase inhibitors, antipsychotics, mood stabilizers, or naltrexone
* in recovery for pathological gambling, due to potential similarity with prize CM, although no increases in gambling have been noted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence based on expired carbon monoxide tests, urinary cotinine tests and self-report. | weeks 5, 12 & 24

SECONDARY OUTCOMES:
Changes from baseline in ambulatory 24-hour systolic blood pressure. | 6 and 24 weeks following the initiation of medication

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Alessi, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States